CLINICAL TRIAL: NCT05311657
Title: Oral Health in Patients With Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Oral Health and Severe COPD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. Antonio Ciardo, Principal Investigator, Heidelberg University
Other Study IDs: S-615/2020
Record Dates: First submitted 2022-03-23; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: COPD; Periodontitis; Caries; Quality of Life; Tooth Loss
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Periodontitis; Tooth Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: Severe COPD (GOLD 3 and 4).
- Control Group: Matched to Test Group regarding age, sex, smoking history and number of systemic diseases.

SUMMARY:
This case-control study aims to investigate the association of severe COPD with oral health.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 40 years and ≤ 85 years;
* Test group: patients with COPD GOLD 3 and 4 with available pulmonary function test values (FEV1, FVC) within the last two weeks;
* Control group: patients without diagnosed or self-suspected pulmonary disease matched for age, sex, smoking and number of systemic diseases to the test group;
* Understanding of measures performed in the study;
* Written informed consent.

Exclusion Criteria:

- Pregnancy.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine pulmonary or dental care.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Tooth loss | one year
  Is the number of teeth different in patients with severe COPD compared to patients without COPD?

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany